CLINICAL TRIAL: NCT03763188
Title: Daily Urinary Urea Excretion to Guide Renal Replacement Therapy Weaning in Intensive Care Units
Brief Title: Dialysis Weaning in Intensive Care Units (Dialysis STOP)
Acronym: D-STOP
Status: Completed | Type: Observational
Sponsor: Dr Alexandre Gros (Individual)
Responsible Party: Sponsor-Investigator, Dr Alexandre Gros, GROS, Alexandre, Medical Doctor, Intensive Care Unit, Principal Investigator, Gros, Alexandre, M.D.
Organization: Gros, Alexandre, M.D. (Individual)
Other Study IDs: AGros
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the group BEFORE: Retrospective group. The daily urinary urea excretion was unknown.
- the group AFTER: Prospective group. Use the daily urinary urea excretion to guide the renal replacement therapy weaning.
  Interventions: Other: Use of daily urinary urea excretion

INTERVENTIONS:
Other: Use of daily urinary urea excretion — Weaning dialysis catheter
  Groups: the group AFTER

SUMMARY:
Evaluation of daily urinary urea excretion, to guide Renal Replacement Therapy weaning, in Intensive Care Units.

The objective is to show that remove the dialysis catheter, once daily urinary urea excretion is greater than 1.35 mmol/kg/d, would increase more than 3 days the number without dialysis catheters, and thus without dialysis, the first 28 days after insertion.

Daily urinary urea excretion = urea (mmol/L) x diuresis (L/d) / weight (kg).

DETAILED DESCRIPTION:
Daily urinary excretion of urea may provide a safe and reproducible renal replacement therapy withdrawal criterion, according to a recent French study (citations). A rate greater than 1.35 mmol/kg/d would predict a weaning success of 97.1% at 1 week. This criterion is influenced by the use of diuretics, and is easily accessible and achievable. Daily urinary urea excretion is representative of the recovery of renal function. The French study establishing this new withdrawal criterion was monocentric and retrospective. However, we changed our practices as soon as we became aware of them.

French multicentric (Bordeaux University Hospital, Libourne, Pau and Bayonne Hospitals) study, before and after:

* Period before: patients who were dialysed in the intensive care units of Bordeaux, Libourne, Pau and Bayonne, from November 2013 to November 2015.
* Period after: patients selected prospectively in the 4 hospitals.

When diuresis > 100 ml/d, an urinary ionogram is realized daily. Measurement of urinary urea excretion every day. Ablation of the catheter as soon as daily urinary urinary excretion > 1.35 mmol/kg/d.

Measurement of daily urinary excretion the following 3 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 of age, who have a Renal Replacement Therapy, in intensive care unit,
* with a diuresis > 100 ml/d.

Exclusion Criteria:

* Patients still presenting "hard" criteria for RRT: metabolic acidosis with pH < 7.15 and PCO2 <50mmHg; acute pulmonary edema (> 5l 02 or 50% FiO2 for Sp02 > 95%) objectified by echocardiography; K> 5.5 mmol/l after treatment
* Renal transplantation
* Long-term chronic kidney injury or short-term dialysis project (arteriovenous fistula created).
* Acute Kidney Injury secondary to thrombotic microangiopathy
* Acute Kidney Injury secondary to an obstacle even if dialysed
* RRT started for toxic cause without IRA (lithium,...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients > 18 years of age, admitted to intensive care unit, who have a RRT for AKI.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
the catheter free days | the first 28 days after catheter insertion
  days

SECONDARY OUTCOMES:
new dialysis catheter and new renal replacement therapy | the first 7 days after dialysis catheter ablation
  number
number of dialysis catheter laid per patients | the first 28 days after catheter insertion
  median
Duration of renal replacement therapy | the first 28 days after catheter insertion
  days
Renal therapy replacement complications (hemorrhage, heparin-induced thrombocytopenia, other) | the first 28 days after catheter insertion
  number
Dialysis catheters infections | the first 28 days after catheter insertion
  number
Duration of ICU stay | the first 28 days after catheter insertion
  days
Duration of mechanical ventilation | the first 28 days after catheter insertion
  days
Mortality at at day 28 | the first 28 days after catheter insertion
  number

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Gros, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aniort J, Ait Hssain A, Pereira B, Coupez E, Pioche PA, Leroy C, Heng AE, Souweine B, Lautrette A. Daily urinary urea excretion to guide intermittent hemodialysis weaning in critically ill patients. Crit Care. 2016 Feb 19;20:43. doi: 10.1186/s13054-016-1225-5. PMID 26895760
- [Derived] Bodot S, Gros A, Le Gall L, Martin A, Gisbert-Mora C, Pillot J, Ragot C, Grand H, Romen A, Masri A, Dewitte A, Gruson D, Prevel R, Rubin S, Orieux A, Boyer A. Effects of the urinary urea excretion index on the decision to wean ICU patients with acute kidney injury from renal replacement therapy: a before-after multicentre study (D-STOP). Crit Care. 2025 Jul 1;29(1):261. doi: 10.1186/s13054-025-05289-8. PMID 40598590